CLINICAL TRIAL: NCT02212483
Title: Clinical Effectiveness and Economical Impact of Medical Indoor Environment Counselors Visiting Homes of Asthma Patients (ECENVIR Study)
Brief Title: Clinical Effectiveness and Economical Impact of Medical Indoor Environment Counselors Visiting Homes of Asthma Patients
Acronym: ECENVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (Other); Institut de Recherche et Documentation en Economie de la Santé, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35RC12_9713_ECENVIR; 2012-A01414-39 (Other: ID RCB); 12/42-875 (Other: CPP); 13.424 (Other: CCTIRS); 913428 (Other: CNIL)
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Asthma; Medical Indoor Environment Counselors; Pediatric; Environment; Clinical effectiveness; Economical impact
MeSH Terms: conditions — Asthma | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Substantial modification of the 20th of June, 2016 : Modification of the design : change into a 2 parallel groups evaluation Justification: At its meeting of June 1, 2016, considering the inclusion difficulties, the Scientific Council decided to give up the "Control" group.
  The study design is then : a prospective multicenter randomised, open label, controlled trial with blind evaluation of the primary evaluation criterion on three parallel groups of patients.
  The objective is to recruit 50 to 70 patients by arm.
  The Control group will still be described.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention group (Experimental): After randomisation and agreement of the patient and the family, the " intervention group " will benefit from a first home intervention of a MIEC during the 4 weeks following inclusion, then a final visit at the end of the study after 12 months.
  Interventions: Other: First home intervention with advice; Other: Final home visit
- Control group (Active Comparator): The " control group " is one of the two comparative groups who will benefit from a first home intervention of a MIEC but without advices (only audit + sampling), then a final and a complete visit at the end of the study.
  This group has been suppressed with the last amendment. But data of the subjects included in this group will be analyzed.
  Interventions: Other: First home intervention without any advice; Other: Final home visit
- Non intervention group (Other): The " non intervention " group is the second comparative group with no initial visit, but will benefit from a complete home intervention of a MIEC at the end of the study.
  Interventions: Other: Final home visit

INTERVENTIONS:
Other: First home intervention with advice — A first home intervention of a MIEC during the 4 weeks following inclusion, with sampling, audit and advices.
  Arms: Intervention group
Other: First home intervention without any advice — A first home intervention of a MIEC during the 4 weeks following inclusion, with sampling, home audit but without any advice.
  Arms: Control group
Other: Final home visit — Final home visit at the end of the study after 12 months, with sampling and home audit.
  For the "intervention group", checking of the advice compliance. For the both comparative groups, delivery of advices.

SUMMARY:
Asthma is one of the most prevalent chronic respiratory diseases, with potential lifethreatening impacts. Indeed, asthma is still responsible for about a thousand deceases per year in France, and constitutes a public health problem in our country as in many countries in the world. The economic burden of asthma is also very high, in terms of health care, and indirect costs including lost work and lost school days.

A few international and French studies have shown a positive clinical impact of Medical Indoor Environment Counselors (MIECs) visiting homes of asthma patients, mainly pediatrics. It has been proposed that MIECs could contribute to reduce patient exposure to many allergens and irritants, among them, house dust mite allergens, formaldehyde or molds. Most of the studies that show a significant decrease of hospitalization or visit in an emergency ward for asthma are monocentric and study the eviction of 1 such identified risk factor. By contrast, meta-analysis underline that additional studies are needed to evaluate the effectiveness of these interventions in adults, in a multicentric and controlled manner, with both clinical, environmental and economical endpoints.

DETAILED DESCRIPTION:
Methodology/Study schedule :

A prospective multicenter randomised, open label, controlled trial with blind evaluation of the primary evaluation criterion on three parallel groups of patients.

Procedures :

Home intervention of MIECs that comprise diagnostic of allergen/irritant exposure (after sampling), advices for allergen/irritant avoidance and follow up of advice compliance.

After randomisation and agreement of the patient and the family, the " intervention group " will benefit from a first home intervention of a MIEC during the 4 weeks following inclusion, then a final visit at the end of the study after 12 months.

Two comparative groups will be identified :

* the " control group " who will benefit from a first home intervention of a MIEC but without advices (only audit + sampling), then a final and a complete visit at the end of the study
* a " non intervention " group with no initial visit, but who will benefit from a complete home intervention of a MIEC at the end of the study.

Substantial modification of the 20th of June, 2016 : Modification of the design : change into a 2 parallel groups evaluation Justification: At its meeting of June 1, 2016, considering the inclusion difficulties, the Scientific Council decided to give up the "Control" group.

The study design is then : a prospective multicenter randomised, open label, controlled trial with blind evaluation of the primary evaluation criterion on three parallel groups of patients.

The objective is to recruit 50 to 70 patients by arm.

Expected findings and impact :

If our hypothesis that home intervention of MIECs are cost-effective on asthma control, then it is relevant to include such service in the medical care during the management of asthma patients with a reimbursement by the social security.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 6 years and less than 45 (<45 years),
* patients with an eligible control level of asthma,
* sensitization to one or more allergens demonstrated during the last 36 months with prick tests (papules with a diameter > 3 mm compared to a negative control or > 50% of positive control) and/or specific IgE detection (> 0.10 U/mL),
* patients > 15 years presenting with a reversibility to ß2-agonists > 200 mL and/or > 12% compared to the initial FEV1 value (test performed at least once in life) or patients ≥ 6 years and ≤ 15 years presenting with a reversibility to ß2-agonists > 200 mL and/or > 12% compared to the initial FEV1 value (at least once in the life) and/or a positive metacholine challenge (at least once in the life),
* patients sleeping > 6 nights per week in the same house
* individuals affiliated to 1 of the 3 French social security (for matching data from French social security via SNIIRAM system),
* Only one patient per dwelling,
* Patient oral consent (written attestation by investigator)

Exclusion Criteria:

* chronic obstructive pulmonary disease (COPD),
* identified occupational asthma,
* Move within the 6 months before home intervention or predicted during the first year of inclusion,
* advices provided during the 2 years before inclusion during a home intervention of a MIEC
* active smokers or smoker who given up smoking less than 5 years ago, with a consumption of more than 10 years of 20 cigarettes/day, OR smoker who given up smoking more than 5 years ago, with a consumption of more than 20 years of 20 cigarettes/day,
* patients < 18 years for whom the parents (or legal guardian) are opposed to the inclusion in ECENVIR study,
* Major people being the object of a legal protection (protection(saving) of justice, guardianship, supervision(guardianship)) and private persons of freedom

Ages: 6 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Therapeutic pressure versus asthma control | 12 months
  The primary objective of this study is to assess the efficacy of home interventions of MIECs on asthma control.

SECONDARY OUTCOMES:
Drug consumption and medical care | 12 months
  One of the secondary objectives is to compare the following after home interventions of MIECs, evolution of drug consumption and medical care needed by asthmatic patients.
Advices compliance | 12 months
  One of the secondary objectives is to compare the following after home interventions of MIECs : compliance with advices of MIECs.
Quality of life questionnaire | 12 months
  One of the secondary objectives is to compare the following after home interventions of MIECs : quality of life before and after home intervention.
Indoor pollutants concentrations | 12 months
  One of the secondary objectives is to compare the following after home interventions of MIECs : evolution of exposure to indoor pollutants in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Gangneux, MD, Principal Investigator — Rennes University Hospital
Locations (16):
- France (16):
  - Strasbourg UH, Strasbourg, Alsace
  - Aix-en-Provence Hospital, Aix-en-Provence
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - Chalon, Chalon-sur-Saône
  - Chauny Hospital, Chauny
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital, Grenoble
  - Lille UH, Lille
  - Marseille European Hospital, Marseille
  - Marseille University Hospital, Marseille
  - Macon Hospital, Mâcon
  - Nantes University Hospital, Nantes
  - Reims University Hospital, Reims
  - Rouen University Hospital, Rouen
  - Vire Hospital, Vire

REFERENCES:
- [Result] Le Cann P, Paulus H, Glorennec P, Le Bot B, Frain S, Gangneux JP. Home Environmental Interventions for the Prevention or Control of Allergic and Respiratory Diseases: What Really Works. J Allergy Clin Immunol Pract. 2017 Jan-Feb;5(1):66-79. doi: 10.1016/j.jaip.2016.07.011. Epub 2016 Sep 21. PMID 27665387
- [Result] Gangneux JP, Bouvrais M, Frain S, Morel H, Deguen S, Chevrier S, Le Cann P. Asthma and Indoor Environment: Usefulness of a Global Allergen Avoidance Method on Asthma Control and Exposure to Molds. Mycopathologia. 2020 Apr;185(2):367-371. doi: 10.1007/s11046-019-00417-9. Epub 2020 Jan 2. PMID 31897973